CLINICAL TRIAL: NCT00648323
Title: A Prospective, Open-Labeled Trial of the Safety and Efficacy of Doxazosin GITS in Patients With Benign Prostate Hyperplasia
Brief Title: Evaluation Of The Efficacy And Safety Of The Doxasozin Gastrointestinal Therapeutic System (GITS) In Patients With Prostate Enlargement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0351063
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Prostate
Keywords: Benign Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Doxazosin mysylate GITS

INTERVENTIONS:
Drug: Doxazosin mysylate GITS — Subjects initiated on 4 mg doxazosin GITS once daily at Visit 1 for four weeks. At Visit 2 (Week 4) increased to 8 mg Doxazosin GITS if efficacy response criteria not met.

SUMMARY:
The primary objectives were to determine the efficacy and safety of the GITS formulation of Doxazosin in Taiwanese patients with prostate enlargement.

ELIGIBILITY:
Inclusion Criteria:

* Taiwanese male subjects between 50 and 80 years of age who had: a primary diagnosis of BPH, defined as having an enlarged prostate (confirmed by digital rectal examination [DRE] and/or B-mode ultrasound); an IPSS score of ≥12; and a Qmax in the range of 5 to 15 mL/sec in a total voided volume of ≥150 mL, were eligible for the study.

Exclusion criteria include but not limited to:

* Previous prostate surgery, presence of a prostate stent or microwave thermotherapy and/or balloon dilatation within the previous 6 months
* Concomitant therapy or previous therapy within 14 days with agents known to affect bladder or urethral function.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-11; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Change in the maximum urinary flow rate (Qmax) from baseline | 8 weeks
Change in the International Prostate Symptom Score (IPSS) total score from baseline | 8 weeks

SECONDARY OUTCOMES:
Change in the International Prostate Symptom Score (IPSS) total score from baseline | 4 weeks
Change in the maximum urinary flow rate (Qmax) from baseline | 4 weeks
Change in the quality of life (QoL) assessment index score from baseline | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Taiwan (4):
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taoyuan District

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0351063&StudyName=Evaluation%20Of%20The%20Efficacy%20And%20Safety%20Of%20The%20Doxasozin%20Gastrointestinal%20Therapeutic%20System%20%28GITS%29%20In%20Patients%20With%20Prostate%20Enlargement